CLINICAL TRIAL: NCT03710252
Title: A Study to Investigate HCV Response Rates in Real World Patients Traditionally Excluded From Clinical Trials: The HEARTLAND Study
Brief Title: A Study to Investigate HCV Response Rates in Real World Patients: HEARTLAND Study
Acronym: HEARTLAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Research Corporation (Network)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLI_IIS_01_2015
Record Dates: First submitted 2018-09-25; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — paritaprevir

STUDY DESIGN:
Intervention Model Description: This is a Phase IV, open label, single arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single (Experimental): Ombitasvir/paritaprevir/ritonavir (OBV/PTV/r) + databuvir (DSV) +/- ribavirin (RBV)
  Interventions: Drug: paritaprevir/ritonavir/ombitasvir + dasabuvir +/- ribavirin

INTERVENTIONS:
Drug: paritaprevir/ritonavir/ombitasvir + dasabuvir +/- ribavirin — OMB/PTV/r + DSV +/- RBV

SUMMARY:
This is a Phase IV, open label, single center study of OBV/PTV/r + DSV +/- RBV for 12 or 24 weeks for the treatment of chronic HCV-1 infection in a real world urban clinical setting.

DETAILED DESCRIPTION:
This is a Phase IV, open label, single center study of OBV/PTV/r + DSV +/- RBV for 12 or 24 weeks for the treatment of chronic HCV-1 infection in a real world urban clinical setting.

The study will enroll chronically infected GT 1 patients who are treatment naïve or who have failed a regimen including pegIFN/RBV +/- telaprevir, boceprevir, or simeprevir.

In addition, up to 20 chronically infected GT1 patients who have traditionally been excluded from clinical trials due to mild to moderate renal insufficiency, irrespective of other co-morbid conditions including poorly controlled diabetes mellitus, high BMI, HIV infection will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * Patients must have chronic GT 1 HCV infection (GT1a, GT1b or GT1a/1b)
  * Patient and partner(s) must agree to use acceptable methods of contraception
  * Patient must be able to read and understand English and/or Spanish
  * Written informed consent

Exclusion Criteria:

* Currently taking or planning on taking any prohibited medications (see US PI)

  * Evidence of decompensated liver disease (Child-Pugh B or C) including the presence of clinical ascites, bleeding varices, or hepatic encephalopathy
  * Abnormal lab values, including:

    * Hemoglobin (Hgb) <8 g/dL
    * Platelets <25,000 cells/mm3
    * Absolute neutrophil count (ANC)<500 cells/mm3
    * Bilirubin >3
    * INR>2.3 ALT/AST > 10 x ULN
    * Serum albumin <2.8
    * GFR <30 mL
  * Alcohol use: >3 drinks per day consistently
  * Uncontrolled HIV or HBV coinfection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The primary analysis will be sustained virologic response 12 weeks after the last treatment dose (SVR12) for the all treated population. | 12 weeks after last treatment
  Primary Analysis

SECONDARY OUTCOMES:
Effect of baseline resistance variants on SVR12 (subgroups: all RAVs, different classes of RAVs) | 12 weeks after last treatment
  Secondary Analysis
Evaluate patient reported outcomes via the SF36v2 survey (subgroups: those who achieve SVR12 and those who do not) | 12 weeks after last treatment
  Secondary Analysis. Comparison between baseline and end of treatment
Evaluate patient adherence (subgroups: those who achieve SVR12 and those who do not) | 12 weeks after last treatment
  Secondary Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fred Poordad, MD, Principal Investigator — American Research Corporation

IPD SHARING:
Plan to Share IPD: Undecided